CLINICAL TRIAL: NCT01944709
Title: Phase I/II Study of Vaccination With Antigen Loaded Dendritic Cells (DCs) in Patients With Inoperable Stage III and Stage IV Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Progressive Disease
Sponsor: Prof. Dr. Silke Gillessen (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Silke Gillessen, lead consultant, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG269/06
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Melanoma
Keywords: melanoma; dendritic cells; peptide; Melan-A
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Dendritic cell application

SUMMARY:
The prognosis of patients with metastatic melanoma is poor and current available treatments are limited. Identification of a number of melanoma-specific tumor antigens that are shared by tumors from different patients, provides attractive targets for immune-based therapies (http://www.bioinfo.org.cn/hptaa/). Different approaches like DNA-/RNA-vaccines, peptide vaccines and dendritic cell (DC) vaccines are under investigation to induce peptide-specific immune responses. In various animal models and in clinical trials it was shown that the most potent induction of anti tumor-specific killer cells was achieved with DC vaccination. DCs are professional antigen presenting cells (APC) that are critical in the initiation of cellular responses in naïve T lymphocytes, in vivo. They are armed with all the molecules needed for the induction of immune responses and have the capacity to migrate into secondary lymphatic organs. In vitro generated dendritic cells are loaded with tumor derived peptides and injected subcutaneously. The concept is to induce or to propagate already existing tumor specific killer T cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma
* Inoperable Stage III or Stage IV melanoma
* Tumor expression of Melan-A and/or NY-Eso-1 by immunohistochemistry
* Human leukocyte antigen (HLA)-A0201 positivity (flow cytometry and PCR)
* Life expectancy more than three months
* Full recovery from surgery
* Karnofsky scale performance status of 70% or more (App II)
* One prior chemo- or cytokine based therapy is allowed
* Age > 18 years
* No uncontrolled infections
* Neutrophile count >1500/ul and thrombocytes >100 000/ul
* Creatinine <1.5 of upper normal level
* Adequate liver function with bilirubin <2 of upper normal level, alanine aminotransferase (ALAT) and aspartate aminotransaminase (ASAT) < 3 x upper normal level
* Clinically significant (i.e. active) cardiovascular disease: Cardiovascular accident (CVA)/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure or serious cardiac arrythmia requiring medication
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient registration, informed consent must be given according to International Conference on Harmonization (ICH)- Good Clinical Practice (GCP), and national/local regulations

Exclusion Criteria:

* Presently clinically significant heart disease (NYHA Class III or IV)
* Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders or uncontrolled peptic ulcer, or seizure or central nervous system disorders
* History of immunodeficiency disease or severe autoimmune disease
* Metastatic disease to the central nervous system
* HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) (test required) or any other severe uncontrolled infection
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry
* Concomitant treatment with steroids or antihistamine drugs. Topical or inhalational steroids are permitted
* Participation in any other clinical trial involving another investigational agent within 6 weeks prior to enrollment
* Pregnancy or lactation
* Women of childbearing potential not using a medically acceptable means of contraception
* Lack of availability of the patient for immunological and clinical follow-up assessment.
* Coagulation or bleeding disorders
* Rapidly progressing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Toxicity as defined by NCI Common Toxicity Criteria Version 3.0 (App I) | 24 hours
  If any grade III or IV toxicity occurs within 24 hours of the vaccine treatment, no further vaccinations will be given. Grade III or IV toxicities arising later will only lead to treatment termination if the toxicity is clinically significant and can be attributed to the vaccination.

SECONDARY OUTCOMES:
Response rates in case of measurable disease | 12 weeks, 20 weeks, 28 weeks
  Three indicator lesions that are measurable in 2 diameters will be assessed radiologically. If there are not three measurable lesions, only the measurable lesions will be assessed.

OTHER OUTCOMES:
Peptide specific cellular immunity: Analyses of peptide specific peripheral blood lymphocytes (PBL) by - tetramer method (flow cytometry) - interferon-gamma ELISPOT | 6 weeks, 12 weeks, 20 weeks, 28 weeks
  Monitoring of immune responses in peripheral blood mononuclear cells (PBMC) via enzyme-linked immunospot (ELISPOT) and Tetramer-staining.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Gillessen, MD, Principal Investigator — Cantonal Hospital St. Gallen, Dept. Oncology
Locations (1):
- Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland